CLINICAL TRIAL: NCT05006612
Title: U/S Guided SAB VS U/S Guided SAB With Modified Pectoral Nerve Block in Modified Radical Mastectomy,Randomized Double Blinded Comparative Study
Brief Title: U/S Guided SAB VS U/S Guided SAB With Modified Pectoral Nerve Block in Modified Radical Mastectomy
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Collaborators: Samuel Bekhet Moawad (Unknown); Ahmed Shaker Ragab (Unknown); Michael Wahib Wadid (Unknown)
Responsible Party: Principal Investigator, Ahmed Abdalla, Professor of Anesthesia &I.C.U and Pain Clinic, Cairo University, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: MS-201-2021
Record Dates: First submitted 2021-07-21; First posted 2021-08-16 (Actual); Last update posted 2022-07-19 (Actual); Status verified 2022-07

CONDITIONS: U/S Guided SAB VS U/S Guided SAB Combined With Modified Pectoral Nerve Block

STUDY DESIGN:
Intervention Model Description: To determine the analgesic effect of ultrasound guided Serratus anterior block combined with modified pectoral nerve block compared to ultrasound guided Serratus Anterior block in patients undergoing modified radical mastectomy regarding the following :
  1-Post-operative opioid (morphine) consumption in the 1st 24 hours 2- Post-operative Numeric Pain Rating Scale.
  3. Effect on hemodynamics:
  Mean arterial blood pressure and Heart rate.
  4. Intraoperative fentanyl consumption.
  5. Duration of analgesic effect
Who Masked: Participant, Investigator
Masking Description: The patients will be randomly assigned into two equal comparable groups using computer- generated random numbers in opaque closed envelopes, each of which will include 30 patients. Randomization will be done by statistician and each group of the patient will revealed only when the included patient is transferred to preanesthetic room.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Group 1 ((Serratus Anterior Plane Block SAPB) (Active Comparator): N=3o Patients will receive Ultrasound guided Serratus Anterior Plane Block with injection of 30 ml levobupivacaine 0.25%.
  Interventions: Procedure: Serratus Anterior Plane Block
- Group 2 ((Serratus Anterior Plane Block SAPB combined with Modified Pectoral Nerve Block) (Active Comparator): N=3o Patients will receive Ultrasound guided Serratus Anterior Plane Block with injection of 20 ml levobupivacaine 0.25%and Modified Pectoral Nerve Block with injection of 10 ml levobupivacaine 0.25%between the two pectoralis muscles, after that, the probe was turned toward the axilla, and as the serratus anterior muscle was recognized above the third and fourth ribs, 10 mL of levobupivacaine 0.25% was injected above this muscle
  Interventions: Procedure: Serratus Anterior Plane Block

INTERVENTIONS:
Procedure: Serratus Anterior Plane Block — SAPB Technique; U/S probe will be placed on the patient's midaxillary line in the transverse plane, at the level of the fifth rib, Then, using U/S guidance, A 38-mm 22-gauge regional block needle is advanced in-plane at an angle of approximately 45 degrees towards the fifth rib. After aspiration to avoid IV injection 30ml of levobupivacaine 0.25% is injected anteriorly to the rib and deep to the serratus anterior muscle.
  SAPB combined with Modified Pectoral Nerve Block :
  SAPB with injection of 20 ml levobupivacaine 0.25% as discussed before. Modified Pectoral Nerve Block:After identification of the axillary vessels, the U/S probe will turned inferolaterally till the serratus anterior and the two pectoralis muscles are detected in one plane. 10 ml of levobupivacaine 0.25%was injected between the two pectoralis muscles. After that,10 mL of levobupivacaine 0.25%is injected above this muscle.
  Other Names: Serratus Anterior Plane Block SAPB combined with Modified Pectoral Nerve Block

SUMMARY:
We hypothesize that ultrasound guided serratus anterior plane block Combined With Modified Pectoral Nerve Block is going to be more effective than Ultrasound guided Serratus anterior plane block alone in patients undergoing MRM as modified Pecs block involves the block of medial and lateral pectoral nerves which are spared in case of serratus block alone, resulting in reducing myofascial pain and opioid consumption.

DETAILED DESCRIPTION:
Ultrasound guided Serratus anterior plane block was introduced in 2013 for analgesia of breast and lateral thoracic wall surgery. At the axillary fossa, the intercostobrachialis nerve, lateral cutaneous branches of the intercostal nerves (T3-T9), long thoracic nerve, and thoracodorsal nerve are located in a compartment between the serratus anterior and the latissimus dorsi muscles, between the posterior and midaxillary lines at this plane local anesthetic will be injected . Complications of serratus anterior plane block include local anesthetic toxicity and pneumothorax , unfortunately medial and lateral pectoral nerves are preserved which are responsible for the myofacial pain .

The pectoral nerves (Pecs) block types I and II (Modified Pectoral block) , is less invasive technique described by Blanco et al where local anesthetic is deposited into the plane between the pectoralis major muscle(PMm) and the pectoralis minor muscle (Pmm) (Pecs I block)and above the serratus anterior muscle at the third rib (Pecs IIblock).,Blocking intercostobrachial, third to sixth intercostals the long thoracic nerves in addition to medial and lateral pectoral nerves.

Addition of Modified Pecs block to Serratus anterior plane block will enhance the control of pain as it block the medial and lateral pectoral nerves which are responsible for the myofacial pain and which are spared in case of Serratus block alone .

ELIGIBILITY:
Inclusion Criteria:

* Female patients
* Type of surgery; Modified Radical Mastectomy (MRM)
* Physical status ASA I, II, III.
* Age ≥ 18 and ≤ 65 Years.
* Body mass index (BMI): > 20 kg/m2 and < 35 kg/m2.

Exclusion Criteria:

* Age <18 years or >65 years
* BMI <20 kg/m2 and >35 kg/m2
* Known sensitivity or contraindication to drug used in the study (local anaesthetics, opioids).
* History of psychological disorders and/or chronic pain.
* Contraindication to regional anaesthesia e.g. local sepsis, pre- existing peripheral neuropathies and coagulopathy.
* Patient refusal.
* Severe respiratory or cardiac disorders.
* Advanced liver or kidney disease.
* Pregnancy.
* Physical status ASA IV and Male patients.

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-06-14 (Actual); Primary Completion 2021-08-16 (Actual); Study Completion 2021-08-23 (Actual)

PRIMARY OUTCOMES:
The total amount of morphine consumption in the first 24 hours postoperatively | Through Study Completion
  The total amount of morphine consumption in the first 24 hours postoperatively

SECONDARY OUTCOMES:
Total amount of intraoperative fentanyl will be recorded. | Through Study Completion over the first 24 hrs postoperative
  Total amount of intraoperative fentanyl will be recorded.
Change in heart rate and mean arterial blood pressure intraoperatively at 30 minutes interval in comparison to baseline reading. | Through Study Completion over the first 24 hrs postoperative
  Change in heart rate and mean arterial blood pressure intraoperatively at 30 minutes interval in comparison to baseline reading.
The degree of postoperative sedation according to Ramsay scores | Through Study Completion over the first 24 hrs postoperative .
  postoperative sedation according to Ramsay scores
Heart rate, mean arterial blood pressure and VAS (at rest and during movement) at 0, 4, 8, 12, 16, 20 and 24 hours postoperatively. | Through Study Completion over the first 24 hrs postoperative
  Change in hemodynamics ((heart rate and mean arterial blood pressure)
Postoperative nausea and vomiting (PONV) as side effects of morphine. | Through Study Completion over the first 24 hrs postoperative
  Nausea and vomiting Scores using a four-point verbal scale:
Time of first rescue analgesia | Through Study Completion over the first 24 hrs postoperative
  Time of first rescue analgesia
Complications related to blocks such as local anaesthetic systemic toxicity, pneumothorax and arterial puncture (US check postoperative). | Through Study Completion over the first 24 hrs postoperative
  Complications related to blocks such as local anaesthetic systemic toxicity, pneumothorax and arterial puncture
Morphine related complications such as respiratory depression, urine retention or pruritis | Through Study Completion over the first 24 hrs postoperative
  Morphine related complications such as respiratory depression, urine retention or pruritis
Patient satisfaction the patient will be classified in this group to satisfied or not. | Through Study Completion over the first 24 hrs postoperative
  Patient satisfaction the patient will be classified in this group to satisfied or not.

CONTACTS AND LOCATIONS:
Locations (1):
- Ahmed Abdalla Mohamed, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: Undecided
Till publication